CLINICAL TRIAL: NCT02801994
Title: Impact of Proportional Assisted Ventilation on Dyspnea and Asynchrony in Mechanically Ventilated Patients
Acronym: DYS-PAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADOREPS_1
Record Dates: First submitted 2016-05-06; First posted 2016-06-16 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Dyspnea
Keywords: Patient-ventilator interaction; Inspiratory muscles; Electromyogram; Mechanical ventilation; Proportional Assist Ventilation
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ventilator settings, PAV (Experimental): A first 30-minutes recording in PSV will be performed. Dyspnea-VAS, IC-RDOS will be measured at the beginning and at the end of this period. EMG and EEG will be recorded continuously. Patients will be subsequently switched to PAV.
  The PAV mode will be delivered by Puritan Bennett 980 ventilator (Covidien, Boulder, USA). Levels of PEEP and FiO2 will be kept constant. The level of assistance in PAV, named %-assistance will be set in order to keep the patient in a respiratory effort zone corresponding to a respiratory muscles pressure time product (PTPmus) between 50 and 150 cm H2O • s / min.
  Interventions: Device: PAV, Puritan Bennett 980 ventilator

INTERVENTIONS:
Device: PAV, Puritan Bennett 980 ventilator — The PAV mode will be delivered by Puritan Bennett 980 ventilator (Covidien, Boulder, USA). Levels of PEEP and FiO2 will be kept constant. The level of assistance in PAV, named %-assistance will be set in order to keep the patient in a respiratory effort zone corresponding to a respiratory muscles pressure time product (PTPmus) between 50 and 150 cm H2O • s / min. As it is not possible to calculate directly the PTPmus at bedside, the investigators will use as a substitute its main component, the pressure peak muscle of the airways according to the previous report from Carteaux et al. This setting has been described extensively and its use has been the subject of a feasibility study in 50 patients. After a 20-minutes stabilization period, a 30-minutes recording will be performed.

SUMMARY:
Rational. The mismatch between the activity of the respiratory muscles and the assistance delivered by the ventilator results in patient-ventilator disharmony, which is commonly observed in ICU patients and is associated with dyspnea and patient-ventilator asynchrony. Both dyspnea and asynchrony are in turn associated with a worse prognosis. Unlike conventional modes of mechanical ventilation, such as pressure support ventilation (PSV) that deliver a constant level of assistance regardless of the patient effort, Proportional Assisted Ventilation (PAV) adjusts the level of ventilator assistance to the activity of respiratory muscles. To date, data on the impact of PAV on dyspnea and patient ventilator asynchrony are scarce and most studies have been conducted in healthy subjects or in ICU patients who had no severe dyspnea nor severe asynchrony. To our knowledge, there are no data in patients with severe patient-ventilator dysharmony.

Study Aim. To evaluate the impact of PAV on dyspnea and patient-ventilator asynchrony in ICU mechanically ventilated patients in intensive care with severe patient-ventilator disharmony defined as either severe dyspnea or severe patient-ventilator asynchrony.

Patients and Methods. Will be included 24 ICU mechanically ventilated patient exhibiting severe patient-ventilator dysharmony with PSV. The intensity of dyspnea will be assessed by the VAS, the ICRDOSS and by the electromyogram of extradiaphragmatic inspiratory muscles and pre inspiratory potential collected from the electroencephalogram. The prevalence of patient-ventilator asynchrony will be quantified.

Expected results. It is anticipated that the switch from PSV to PAV will decrease the prevalence and severity of dyspnea and the prevalence of patient-ventilator asynchrony.

DETAILED DESCRIPTION:
Rational As opposed to controlled mechanical ventilation, partial modes of assisted ventilation maintains a certain level spontaneous activity of respiratory muscles. As a consequence, assisted ventilation may contribute to prevents ventilator induced diaphragm dysfunction (1-3), improves gas exchanges (4), reduces the use of sedative agents, which can ultimately shorten weaning from mechanical ventilation (5).

The most widely used partial ventilatory assistance mode is pressure support ventilation (PSV) (6), in which a constant preset level of pressure assists each inspiration regardless of the patient's inspiratory effort. Mismatching between patient demand and level of assistance, which the investigators will term patient-ventilator dysharmony in the present project is therefore possible and can be potentially harmful. On the one hand, underassistance may induce respiratory discomfort and dyspnea (7), which is an immediate cause of suffering, generates anxiety and is a source of delayed neuropsychological sequelae such as dark respiratory recollections and post-traumatic stress disorders(8-12). One the other hand, overassistance may cause lung overdistension and volutrauma (13). Finally, both underassistance and overassistance may generate patient-ventilator asynchrony that is associated with poorer clinical outcomes (14). Of notice, underassistance is likely to be associated with an asynchrony named double-triggering while over assistance is more commonly associated with ineffective efforts(15).

Proportional modes of mechanical ventilation have been designed to overcome this weakness of (PSV). Indeed, as opposed to PSV that delivers a constant level of assistance regardless of the patient inspiratory effort, proportional modes of ventilation adjust the amount of assistance delivered with respect to the patient's efforts. Proportional Assisted Ventilation (PAV) is one of these modes and adjusts ventilator assistance to the activity of respiratory muscles estimated by an algorithm (16-23). Previous studies have shown the potential benefits of PAV to prevent the risk of overassistance(24) and in turn to reduce the prevalence of ineffective effort (25-28). In addition, PAV increases the variability of the breathing pattern (17, 20-23, 29-32). To date, data on the impact of PAV on dyspnea and patient ventilator asynchrony are scarce (24-28, 33). Most of these works have been conducted in healthy subjects or in ICU patients with no severe dyspnea nor severe asynchrony (24-28, 33). To our knowledge, there are no data in patients with severe patient-ventilator dysharmony.

Because PAV adjusts the level of assistance to the activity of respiratory muscles, a surrogate of the respiratory drive, it is licit to hypothesize that PAV should prevent severe patient-ventilator dysharmony, defined as either severe dyspnea or severe patient-ventilator asynchrony.

The objective of the present research proposal is to evaluate the impact of PAV on dyspnea and patient-ventilator asynchrony in ICU mechanically ventilated patients in intensive care with severe patient-ventilator disharmony defined as either severe dyspnea or severe patient-ventilator asynchrony.

The specific objectives are to compare in these patients the impact of a switch of the ventilator mode from PSV to PAV in terms of:

1. The intensity of dyspnea quantified by a self-assessment visual analogic scale and by two electrophysiological tools such as the electromyogram of extradiaphragmatic inspiratory muscles and the pre inspiratory potentials on the electroencephalogram (see below, Patients and Methods).
2. The prevalence of two major patient-ventilator asynchronies that are ineffective efforts and double triggering (see below, Patients and Methods).

Materials and methods used and statistical methods

This observational, single-centre prospective study will be performed in the Medical intensive care unit (ICU) of the Respiratory and ICU Division of Pitié-Salpêtrière hospital, Paris, France.

1. Population, sampling The inclusion of patients will be done after informing patients and obtaining their informed consent.

1.1 Inclusion criteria Patients will be included as soon as the meet the following criteria.

* Intubation and mechanical ventilation for a respiratory cause with severe hypoxemia defined as a PaO2 to FiO2 ratio <300 recorded at least once during the present ICU stay.
* PSV ventilation for > 6 hours.
* Severe patient-ventilator disharmony
* Decision of the physician in charge of the patient to switch mechanical ventilation from PSV mode to PAV.
* Remaining duration of mechanical ventilation estimated ≥ 24 hours. 1.2 Exclusion criteria Exclusion criteria will be as follows.
* Severe hypoxemia defined as a PaO2 to FiO2 ratio <150 mmHg.
* Delirium according to the CAM-ICU (1)
* Hemodynamic instability defined by the need for intravenous fluids or catecholamine during the previous 24 hours.
* Age <18 years; pregnant woman. 1.3 sample size Our objective is to study a convenient sample of 24 patients. Given the recruitment unit, the duration of the study should be 6 months.

  2 Study design A first 10-minutes recording in PSV will be performed. Dyspnea-VAS, IC-RDOS will be measured at the beginning and at the end of this period. EMG and EEG will be recorded continuously. Patients will be subsequently switched to PAV.

The PAV mode will be delivered by Puritan Bennett 980 ventilator (Covidien, Boulder, USA). Levels of PEEP and FiO2 will be kept constant. The level of assistance in PAV, named %-assistance will be set in order to keep the patient in a respiratory effort zone corresponding to a respiratory muscles pressure time product (PTPmus) between 50 and 150 cm H2O • s / min (8). As it is not possible to calculate directly the PTPmus at bedside, the investigators will use as a substitute its main component, the pressure peak muscle of the airways according to the previous report from Carteaux et al.(8). This setting has been described extensively and its use has been the subject of a feasibility study in 50 patients. After a 10-minutes stabilization period, a 10-minutes recording will be performed. Dyspnea-VAS, IC-RDOS will be measured at the beginning and at the end of this period. EMG and EEG will be recorded continuously.

During the whole procedure, the usual hemodynamic and respiratory variables - non-invasive blood pressure or invasive if any, pulse oximetry, respiratory rate, - will be monitored continuously.

4 Statistical analysis Statistical analysis will be conducted with the Prism 5.0 software (GraphPad Software, USA). The distribution followed by the analysed data will be evaluated by the normality test of Kolmogorov-Smirnov. Probability of Type I error p less than or equal to 0.05 will be considered statistically significant. To investigate the effects of ventilation mode, the descriptors of dyspnea, the amplitude of the EMG as well as the PPI will be compared using a Mann-Whitney test. The prevalence of main asynchronies will be compared with a

ELIGIBILITY:
Inclusion Criteria:

Patients will be included as soon as the meet the following criteria.

* Intubation and mechanical ventilation for a respiratory cause with severe hypoxemia defined as a PaO2 to FiO2 ratio <300 recorded at least once during the present ICU stay.
* PSV ventilation for > 6 hours.
* Severe patient-ventilator disharmony defined by either

  * a dyspnea ≥ 4 on a visual analogic scale (VAS) from 0 to 10 with respiratory rate ≥ 24 /minute and a drawing of neck muscles,
  * or by an asynchrony index (IA) ≥ 10%, defined as = number of asynchrony events/total respiratory rate (ventilator cycles +wasted efforts) × 100
* No improvement of disharmony despite an optimization of ventilator setting defined as follows.

  * No improvement of dyspnea or double triggering despite an increase of the level of pressure support that should not generate a tidal volume > 10 ml/kg
  * No improvement of ineffective efforts despite a decrease of the level of pressure support or generation of a dyspnea (defined as VAS>4) in response of the decrease of the level of pressure support.
* Decision of the physician in charge of the patient to switch mechanical ventilation from PSV mode to PAV.
* Remaining duration of mechanical ventilation estimated ≥ 24 hours.
* Patient able to communicate (Richmond Agitation and Sedation Scale between -1 and +1).

Exclusion Criteria:

* Exclusion criteria will be as follows.

  * Severe hypoxemia defined as a PaO2 to FiO2 ratio <150 mmHg.
  * Delirium according to the CAM-ICU (1)
  * Hemodynamic instability defined by the need for intravenous fluids or catecholamine during the previous 24 hours.
  * Age <18 years; pregnant woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Quantification of dyspnea | in real time, during the procedure
  Dyspnea will be quantified with with the ICU Respiratory Distress Operating Scale (IC-RDOS)

SECONDARY OUTCOMES:
Airway pressure | in real time, during the procedure
  The airway pressure will be also measured at the Y-piece by a differential pressure transducer (Validyne, Northridge, USA).
Electromyography (EMG) of extra inspiratory diaphragmatic muscles | in real time, during the procedure
  The amplitude of the EMG signal of extradiaphragmatics inspiratory muscles is proportional to the intensity of dyspnea. EMG will be collected by self-adhesive surface electrodes of the same type as those commonly used to collect the ECG signal in critically ill patients. A distance of 2 cm will separate the two electrodes. The position of the electrodes will depend on the recorded muscle.
Electroencephalogram (EEG) in search of a pre-inspiratory potential | in real time, during the procedure
  The application of an inspiratory resistive load to healthy subjects results in the activation of the pre-motor cortex detected by EEG recording. This EEG activity is named pre-inspiratory potential (PIP).
Arterial blood gas | in real time, during the procedure
  For patients with an arterial catheter, the measurement of blood gases using an arterial blood sample of a volume of less than 1ml be performed at the end of each condition.
Patient-ventilator asynchrony | in real time, during the procedure
  Asynchrony will be detected by visual inspection of the recordings. The investigators will investigate patterns of two major asynchronies that are easily detected on pressure and flow recordings: ineffective triggering and double triggering. Ineffective triggering will be defined as an abrupt airway pressure drop (≥ 0.5 cmH2O) simultaneous to a flow decrease (in absolute value) and not followed by an assisted cycle during the expiratory period. Double-triggering will be defined as two cycles separated by a very short expiratory time, defined as less than one-half of the mean inspiratory time, the first cycle being patient-triggered.
Flow | in real time, during the procedure
  Airway flow will be measured with a pneumotachograph (Hans Rudolph, Kansas City, USA) inserted between the Y-piece and the endotracheal tube and connected to a differential pressure sensor (Validyne, Northridge, USA).
Quantification of dyspnea | in real time, during the procedure
  Dyspnea will be quantified with a dyspnea-VAS from 0 (no discomfort) to 10 (maximum breathing)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pneumologie et Réanimation Médicale, Groupe Hospitalier Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Result] Campbell ML. Psychometric testing of a respiratory distress observation scale. J Palliat Med. 2008 Jan-Feb;11(1):44-50. doi: 10.1089/jpm.2007.0090. PMID 18370892
- [Result] Campbell ML, Templin T, Walch J. A Respiratory Distress Observation Scale for patients unable to self-report dyspnea. J Palliat Med. 2010 Mar;13(3):285-90. doi: 10.1089/jpm.2009.0229. PMID 20078243
- [Result] Raux M, Ray P, Prella M, Duguet A, Demoule A, Similowski T. Cerebral cortex activation during experimentally induced ventilator fighting in normal humans receiving noninvasive mechanical ventilation. Anesthesiology. 2007 Nov;107(5):746-55. doi: 10.1097/01.anes.0000287005.58761.e8. PMID 18073550
- [Result] Raux M, Straus C, Redolfi S, Morelot-Panzini C, Couturier A, Hug F, Similowski T. Electroencephalographic evidence for pre-motor cortex activation during inspiratory loading in humans. J Physiol. 2007 Jan 15;578(Pt 2):569-78. doi: 10.1113/jphysiol.2006.120246. Epub 2006 Nov 16. PMID 17110415
- [Result] Carteaux G, Mancebo J, Mercat A, Dellamonica J, Richard JC, Aguirre-Bermeo H, Kouatchet A, Beduneau G, Thille AW, Brochard L. Bedside adjustment of proportional assist ventilation to target a predefined range of respiratory effort. Crit Care Med. 2013 Sep;41(9):2125-32. doi: 10.1097/CCM.0b013e31828a42e5. PMID 23787397
- [Result] Thille AW, Rodriguez P, Cabello B, Lellouche F, Brochard L. Patient-ventilator asynchrony during assisted mechanical ventilation. Intensive Care Med. 2006 Oct;32(10):1515-22. doi: 10.1007/s00134-006-0301-8. Epub 2006 Aug 1. PMID 16896854
- [Result] Dres M, Schmidt M, Ferre A, Mayaux J, Similowski T, Demoule A. Diaphragm electromyographic activity as a predictor of weaning failure. Intensive Care Med. 2012 Dec;38(12):2017-25. doi: 10.1007/s00134-012-2700-3. Epub 2012 Sep 26. PMID 23011532
- [Result] Hug F, Raux M, Morelot-Panzini C, Similowski T. Surface EMG to assess and quantify upper airway dilators activity during non-invasive ventilation. Respir Physiol Neurobiol. 2011 Sep 15;178(2):341-5. doi: 10.1016/j.resp.2011.06.007. Epub 2011 Jun 15. PMID 21699998
- [Result] Schmidt M, Chiti L, Hug F, Demoule A, Similowski T. Surface electromyogram of inspiratory muscles: a possible routine monitoring tool in the intensive care unit. Br J Anaesth. 2011 Jun;106(6):913-4. doi: 10.1093/bja/aer141. No abstract available. PMID 21576107
- [Result] Schmidt M, Kindler F, Gottfried SB, Raux M, Hug F, Similowski T, Demoule A. Dyspnea and surface inspiratory electromyograms in mechanically ventilated patients. Intensive Care Med. 2013 Aug;39(8):1368-76. doi: 10.1007/s00134-013-2910-3. Epub 2013 Apr 11. PMID 23575612
- [Result] Gayan-Ramirez G, Testelmans D, Maes K, Racz GZ, Cadot P, Zador E, Wuytack F, Decramer M. Intermittent spontaneous breathing protects the rat diaphragm from mechanical ventilation effects. Crit Care Med. 2005 Dec;33(12):2804-9. doi: 10.1097/01.ccm.0000191250.32988.a3. PMID 16352963
- [Result] Sassoon CS, Zhu E, Caiozzo VJ. Assist-control mechanical ventilation attenuates ventilator-induced diaphragmatic dysfunction. Am J Respir Crit Care Med. 2004 Sep 15;170(6):626-32. doi: 10.1164/rccm.200401-042OC. Epub 2004 Jun 16. PMID 15201132
- [Result] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Result] Putensen C, Zech S, Wrigge H, Zinserling J, Stuber F, Von Spiegel T, Mutz N. Long-term effects of spontaneous breathing during ventilatory support in patients with acute lung injury. Am J Respir Crit Care Med. 2001 Jul 1;164(1):43-9. doi: 10.1164/ajrccm.164.1.2001078. PMID 11435237
- [Result] Brochard L, Rauss A, Benito S, Conti G, Mancebo J, Rekik N, Gasparetto A, Lemaire F. Comparison of three methods of gradual withdrawal from ventilatory support during weaning from mechanical ventilation. Am J Respir Crit Care Med. 1994 Oct;150(4):896-903. doi: 10.1164/ajrccm.150.4.7921460.
- [Result] Esteban A, Ferguson ND, Meade MO, Frutos-Vivar F, Apezteguia C, Brochard L, Raymondos K, Nin N, Hurtado J, Tomicic V, Gonzalez M, Elizalde J, Nightingale P, Abroug F, Pelosi P, Arabi Y, Moreno R, Jibaja M, D'Empaire G, Sandi F, Matamis D, Montanez AM, Anzueto A; VENTILA Group. Evolution of mechanical ventilation in response to clinical research. Am J Respir Crit Care Med. 2008 Jan 15;177(2):170-7. doi: 10.1164/rccm.200706-893OC. Epub 2007 Oct 25. PMID 17962636
- [Result] Schmidt M, Banzett RB, Raux M, Morelot-Panzini C, Dangers L, Similowski T, Demoule A. Unrecognized suffering in the ICU: addressing dyspnea in mechanically ventilated patients. Intensive Care Med. 2014 Jan;40(1):1-10. doi: 10.1007/s00134-013-3117-3. Epub 2013 Oct 17. PMID 24132382
- [Result] Schmidt M, Demoule A, Polito A, Porchet R, Aboab J, Siami S, Morelot-Panzini C, Similowski T, Sharshar T. Dyspnea in mechanically ventilated critically ill patients. Crit Care Med. 2011 Sep;39(9):2059-65. doi: 10.1097/CCM.0b013e31821e8779. PMID 21572329
- [Result] de Miranda S, Pochard F, Chaize M, Megarbane B, Cuvelier A, Bele N, Gonzalez-Bermejo J, Aboab J, Lautrette A, Lemiale V, Roche N, Thirion M, Chevret S, Schlemmer B, Similowski T, Azoulay E. Postintensive care unit psychological burden in patients with chronic obstructive pulmonary disease and informal caregivers: A multicenter study. Crit Care Med. 2011 Jan;39(1):112-8. doi: 10.1097/CCM.0b013e3181feb824. PMID 21037472
- [Result] Rotondi AJ, Chelluri L, Sirio C, Mendelsohn A, Schulz R, Belle S, Im K, Donahoe M, Pinsky MR. Patients' recollections of stressful experiences while receiving prolonged mechanical ventilation in an intensive care unit. Crit Care Med. 2002 Apr;30(4):746-52. doi: 10.1097/00003246-200204000-00004. PMID 11940739
- [Result] Pochard F, Lanore JJ, Bellivier F, Ferrand I, Mira JP, Belghith M, Brunet F, Dhainaut JF. Subjective psychological status of severely ill patients discharged from mechanical ventilation. Clin Intensive Care. 1995;6(2):57-61. PMID 10150800
- [Result] Cuthbertson BH, Hull A, Strachan M, Scott J. Post-traumatic stress disorder after critical illness requiring general intensive care. Intensive Care Med. 2004 Mar;30(3):450-5. doi: 10.1007/s00134-003-2004-8. Epub 2003 Sep 5. PMID 12961065
- [Result] Dreyfuss D, Soler P, Basset G, Saumon G. High inflation pressure pulmonary edema. Respective effects of high airway pressure, high tidal volume, and positive end-expiratory pressure. Am Rev Respir Dis. 1988 May;137(5):1159-64. doi: 10.1164/ajrccm/137.5.1159. PMID 3057957
- [Result] Alexopoulou C, Kondili E, Plataki M, Georgopoulos D. Patient-ventilator synchrony and sleep quality with proportional assist and pressure support ventilation. Intensive Care Med. 2013 Jun;39(6):1040-7. doi: 10.1007/s00134-013-2850-y. Epub 2013 Feb 16. PMID 23417203
- [Result] Younes M, Webster K, Kun J, Roberts D, Masiowski B. A method for measuring passive elastance during proportional assist ventilation. Am J Respir Crit Care Med. 2001 Jul 1;164(1):50-60. doi: 10.1164/ajrccm.164.1.2010068. PMID 11435238
- [Result] Younes M, Kun J, Masiowski B, Webster K, Roberts D. A method for noninvasive determination of inspiratory resistance during proportional assist ventilation. Am J Respir Crit Care Med. 2001 Mar;163(4):829-39. doi: 10.1164/ajrccm.163.4.2005063. PMID 11282753
- [Result] Younes M, Puddy A, Roberts D, Light RB, Quesada A, Taylor K, Oppenheimer L, Cramp H. Proportional assist ventilation. Results of an initial clinical trial. Am Rev Respir Dis. 1992 Jan;145(1):121-9. doi: 10.1164/ajrccm/145.1.121. PMID 1731574
- [Result] Younes M. Proportional assist ventilation, a new approach to ventilatory support. Theory. Am Rev Respir Dis. 1992 Jan;145(1):114-20. doi: 10.1164/ajrccm/145.1.114. PMID 1731573
- [Result] Wysocki M, Meshaka P, Richard JC, Similowski T. Proportional-assist ventilation compared with pressure-support ventilation during exercise in volunteers with external thoracic restriction. Crit Care Med. 2004 Feb;32(2):409-14. doi: 10.1097/01.CCM.0000108869.12426.51. PMID 14758156
- [Result] Ranieri VM, Giuliani R, Mascia L, Grasso S, Petruzzelli V, Puntillo N, Perchiazzi G, Fiore T, Brienza A. Patient-ventilator interaction during acute hypercapnia: pressure-support vs. proportional-assist ventilation. J Appl Physiol (1985). 1996 Jul;81(1):426-36. doi: 10.1152/jappl.1996.81.1.426. PMID 8828695
- [Result] Grasso S, Puntillo F, Mascia L, Ancona G, Fiore T, Bruno F, Slutsky AS, Ranieri VM. Compensation for increase in respiratory workload during mechanical ventilation. Pressure-support versus proportional-assist ventilation. Am J Respir Crit Care Med. 2000 Mar;161(3 Pt 1):819-26. doi: 10.1164/ajrccm.161.3.9902065. PMID 10712328
- [Result] Kondili E, Prinianakis G, Alexopoulou C, Vakouti E, Klimathianaki M, Georgopoulos D. Respiratory load compensation during mechanical ventilation--proportional assist ventilation with load-adjustable gain factors versus pressure support. Intensive Care Med. 2006 May;32(5):692-9. doi: 10.1007/s00134-006-0110-0. Epub 2006 Mar 8. PMID 16523329
- [Result] Giannouli E, Webster K, Roberts D, Younes M. Response of ventilator-dependent patients to different levels of pressure support and proportional assist. Am J Respir Crit Care Med. 1999 Jun;159(6):1716-25. doi: 10.1164/ajrccm.159.6.9704025. PMID 10351909
- [Result] Appendini L, Purro A, Gudjonsdottir M, Baderna P, Patessio A, Zanaboni S, Donner CF, Rossi A. Physiologic response of ventilator-dependent patients with chronic obstructive pulmonary disease to proportional assist ventilation and continuous positive airway pressure. Am J Respir Crit Care Med. 1999 May;159(5 Pt 1):1510-7. doi: 10.1164/ajrccm.159.5.9804130. PMID 10228119
- [Result] Passam F, Hoing S, Prinianakis G, Siafakas N, Milic-Emili J, Georgopoulos D. Effect of different levels of pressure support and proportional assist ventilation on breathing pattern, work of breathing and gas exchange in mechanically ventilated hypercapnic COPD patients with acute respiratory failure. Respiration. 2003 Jul-Aug;70(4):355-61. doi: 10.1159/000072897. PMID 14512669
- [Result] Xirouchaki N, Kondili E, Vaporidi K, Xirouchakis G, Klimathianaki M, Gavriilidis G, Alexandopoulou E, Plataki M, Alexopoulou C, Georgopoulos D. Proportional assist ventilation with load-adjustable gain factors in critically ill patients: comparison with pressure support. Intensive Care Med. 2008 Nov;34(11):2026-34. doi: 10.1007/s00134-008-1209-2. Epub 2008 Jul 8. PMID 18607562
- [Result] Bosma K, Ferreyra G, Ambrogio C, Pasero D, Mirabella L, Braghiroli A, Appendini L, Mascia L, Ranieri VM. Patient-ventilator interaction and sleep in mechanically ventilated patients: pressure support versus proportional assist ventilation. Crit Care Med. 2007 Apr;35(4):1048-54. doi: 10.1097/01.CCM.0000260055.64235.7C. PMID 17334259
- [Result] Fernandez-Vivas M, Caturla-Such J, Gonzalez de la Rosa J, Acosta-Escribano J, Alvarez-Sanchez B, Canovas-Robles J. Noninvasive pressure support versus proportional assist ventilation in acute respiratory failure. Intensive Care Med. 2003 Jul;29(7):1126-33. doi: 10.1007/s00134-003-1768-1. Epub 2003 Jun 12. PMID 12802487
- [Result] Gay PC, Hess DR, Hill NS. Noninvasive proportional assist ventilation for acute respiratory insufficiency. Comparison with pressure support ventilation. Am J Respir Crit Care Med. 2001 Nov 1;164(9):1606-11. doi: 10.1164/ajrccm.164.9.2011119. PMID 11719297
- [Result] Hernandez P, Maltais F, Gursahaney A, Leblanc P, Gottfried SB. Proportional assist ventilation may improve exercise performance in severe chronic obstructive pulmonary disease. J Cardiopulm Rehabil. 2001 May-Jun;21(3):135-42. doi: 10.1097/00008483-200105000-00003. PMID 11409222
- [Result] Wysocki M, Richard JC, Meshaka P. Noninvasive proportional assist ventilation compared with noninvasive pressure support ventilation in hypercapnic acute respiratory failure. Crit Care Med. 2002 Feb;30(2):323-9. doi: 10.1097/00003246-200202000-00010. PMID 11889302
- [Result] Mols G, von Ungern-Sternberg B, Rohr E, Haberthur C, Geiger K, Guttmann J. Respiratory comfort and breathing pattern during volume proportional assist ventilation and pressure support ventilation: a study on volunteers with artificially reduced compliance. Crit Care Med. 2000 Jun;28(6):1940-6. doi: 10.1097/00003246-200006000-00042. PMID 10890645